CLINICAL TRIAL: NCT00594516
Title: A Randomized, Double-Blind, 2-Period, Crossover Study to Establish the Dose Equivalence and Direct Conversion Between Immediate Release (IR) and Extended-Release (ER) CG5503 in Subjects With Moderate-to-Severe, Chronic Low Back Pain
Brief Title: Study on the Safety and Effectiveness of Switching Between Two Forms of Tapentadol in Patients With Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Director, Clinical Leader, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CR014242; R331333PAI3019
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Results first posted 2010-07-26 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Dose Equivalence; Tapentadol (CG5503); Tapentadol-IR; Tapentadol-ER
MeSH Terms: conditions — Low Back Pain | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 001 (Experimental): tapentadol (CG5503) Immediate Release (IR) Following open label period is 2 double blind periods: Tapentadol IR in first intervention period of double-blind phase and Tapentadol ER 100 150 200 or 250 mg tablets twice daily in second or Tapentadol ER in first intervention period of double-blind phase and Tapentadol IR in second,tapentadol (CG5503) Immediate Release IR 21 day Open Label: an adjustable dose of Tapentadol IR 50-100mg orally every 4-6 hours to maximum total daily dose (TDD) dose of 500 mg during open label period
  Interventions: Drug: tapentadol (CG5503) Immediate Release IR; Drug: tapentadol (CG5503) Immediate Release (IR)
- 002 (Experimental): tapentadol (CG5503) Extended Release (ER) During 2 double blind periods: Tapentadol ER 100 150 200 or 250 mg tablets twice daily in the first intervention period of double-blind phase and Tapentadol IR in the second or Tapentadol IR in first intervention period of double-blind phase and Tapentadol ER in second
  Interventions: Drug: tapentadol (CG5503) Extended Release (ER)

INTERVENTIONS:
Drug: tapentadol (CG5503) Immediate Release IR — 21 day Open Label: an adjustable dose of Tapentadol IR 50-100mg orally every 4-6 hours to maximum total daily dose (TDD) dose of 500 mg during open label period
  Arms: 001
Drug: tapentadol (CG5503) Extended Release (ER) — During 2 double blind periods: Tapentadol ER 100, 150, 200 or 250 mg tablets twice daily in the first intervention period of double-blind phase and Tapentadol IR in the second or Tapentadol IR in first intervention period of double-blind phase and Tapentadol ER in second
  Arms: 002
Drug: tapentadol (CG5503) Immediate Release (IR) — Following open label period is 2 double blind periods: Tapentadol IR in first intervention period of double-blind phase and Tapentadol ER 100, 150, 200 or 250 mg tablets twice daily in second or Tapentadol ER in first intervention period of double-blind phase and Tapentadol IR in second
  Arms: 001

SUMMARY:
The objective of this study is to test the idea that the immediate-release (IR) form of tapentadol (CG5503) can be directly converted into an approximately equivalent total daily dose (TDD) of the extended-release (ER) form, and vice-versa, with equivalent safety and efficacy.

DETAILED DESCRIPTION:
This study will establish the dose equivalence and the safety and effectiveness of the Immediate Release (IR) and Extended Release (ER) forms of tapentadol (CG5503) to support the conversion from IR to ER, and ER to IR use. Dose equivalence will be examined in patients diagnosed with moderate-to-severe, chronic Low Back Pain (LBP) requiring drug treatment for at least 3 months, and who are dissatisfied with current therapy. The study consists of 5 periods: a screening period during which patients are evaluated for study eligibility; a 21-day open-label period to find the best, stable dose of tapentadol (CG5503) IR for each patient individually; a 14-day double-blind period when patients are randomly chosen either to continue for 14 days on the stable IR dose from the open-label period or switch to the ER form; a second, 14-day period during which patients switch to whichever form of tapentadol (CG5503) they did not take during the first 14-day period (the total daily dose [TDD] remains approximately equivalent for the IR and ER forms throughout both double-blind periods); and a follow-up period. During the study, pain levels will be recorded and overall safety measures taken. The expectation (thought) is that approximately equivalent doses of both forms of tapentadol (CG5503) provide equivalent effectiveness and safety and that the two forms can be directly converted by dividing the total daily dose by the number of times the drug is taken each day. During the 21-day open-label period, 50, 75 or 100mg of the IR form is given orally every 4 or 6 hours, starting with 50mg every 6 hours. Then, the dose, the frequency of giving the drug, or both may be increased, to a maximum TDD of 500mg, or decreased in 50 mg increments, with minimum TDD of 200 mg, until the optimal stable dose for a patient is found. During the 2 double-blind periods, a TDD approximately equivalent to the stable open-label dose is given orally in IR (or ER) form or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Low Back Pain (LBP) of non-malignant origin present for at least 3 months immediately before study entry
* Taking drug treatment for pain for at least 3 months before screening and who are dissatisfied with current therapy
* Subjects receiving opioid treatment must have a total daily opioid dose <= 160 mg/day of oral morphine equivalent
* For entry into open label period patients must have a baseline score >=5 on an 11-point NRS, calculated as the average pain intensity during the last 3 days of the washout period
* For entry into the double-blind period subjects must have remained on the same optimal stable dose and frequency of tapentadol (CG5503) IR administration during the last 3 days of the open-label treatment period

Exclusion Criteria:

* Presence of conditions other than Low Back Pain (LBP) that could make it hard to assess or self-evaluate pain
* Surgery in low back area within 3 months of screening or expected surgery in the low back area during the study
* Any scheduled surgery or painful procedure during the study, or any clinically significant disease that, in the opinion of the investigator, may affect efficacy or safety assessments
* History of malignancy within the past 2 years, with the exception of basal cell carcinoma that has been treated and is no longer present
* Women who are pregnant or breast-feeding
* Moderately or severely impaired liver function
* Severely impaired kidney function
* History of chronic hepatitis B or C, or HIV, or presence of active hepatitis B or C in past 3 months
* History of seizure disorder
* Alcohol or drug abuse
* Uncontrolled high blood pressure
* Clinically relevant history of hypersensitivity, allergy, or contraindications to acetaminophen or opioid analgesics (or ingredients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-12; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Etropolski MS, Okamoto A, Shapiro DY, Rauschkolb C. Dose conversion between tapentadol immediate and extended release for low back pain. Pain Physician. 2010 Jan-Feb;13(1):61-70. PMID 20119464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first site opened on 30 November 2007. The recruitment period for this outpatient, multicenter study occurred between 10 December 2007 and 01 May 2008.
Pre-assignment Details: The study consisted of screening period (up to 21 days), washout period (from 3 to 7 days), open label (OL) treatment period (3 weeks), followed by a double blind (DB) active treatment period, with crossover design of 2 randomized sequences of tapentadol immediate release (IR) to tapentadol extended release (ER) and tapentadol ER to IR (4 weeks)
Groups:
- Tapentadol: Subjects treated in the Tapentadol(CG5503) Immediate Release (IR) Open-Label period
- Tapentadol IR to ER: Tapentadol IR in first intervention period of double-blind phase and Tapentadol ER in second intervention period of double-blind phase
- Tapentadol ER to IR: Tapentadol ER in first intervention period of double-blind phase and Tapentadol IR in second intervention period of double-blind phase
Period: Open Label (OL): Tapentadol IR
Arm/Group | Tapentadol | Tapentadol IR to ER | Tapentadol ER to IR
Started | 116 (one patient was enrolled but lost to follow up at the start of open label therefore was not included) | 0 | 0
Completed | 87 | 0 | 0
Not Completed | 29 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Adverse Event | 16 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Study Medication Non Compliant | 6 | 0 | 0
Period: DB: Tapentadol IR to ER & ER to IR
Arm/Group | Tapentadol | Tapentadol IR to ER | Tapentadol ER to IR
Started | 0 | 44 | 43
Completed | 0 | 37 | 35
Not Completed | 0 | 7 | 8
Not completed — Withdrawal by Subject | 0 | 3 | 3
Not completed — Study Medication Non compliant | 0 | 3 | 2
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tapentadol
Number analyzed (Participants) | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 86
  >=65 years | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (15.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 51
Race/Ethnicity, Customized [Number; unit: participants] — Race/ethnicity
  participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 14
    White | 90
    Hispanic or Latino | 12
    Other | 0

OUTCOME MEASURES:

1. Primary Outcome: The Difference in the Mean Average Pain Intensity Score on an 11-point Numerical Rating Scale (NRS) During the Last 3 Days of Each Double-blind Treatment Period. (Difference Between Two DB Randomization Treatment Sequences)
Description: For this twice daily pain assessment, the subjects were to indicate the level of average pain experienced over the previous 12 hours on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: 14 days for each cross-over period
Population: Per-protocol set defined as the number of randomized subjects who took at least one dose of study drug during the DB treatment period, and who met additional criteria which were identified prior to unblinding.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Tapentadol: Subjects treated in the Tapentadol Immediate Release (IR) Open-Label period (followed by randomization to double-blind crossover maintenance period in which all subjects receive both IR and ER formulations)
Arm/Group | Tapentadol
Number analyzed (Participants) | 60
Units on a scale | 0.1 [-0.09 to 0.28]
Statistical Analysis 1: Comparison: Tapentadol; Comparison of Tapentadol IR to ER analysis of variance model with factors for treatment, double blind cross-over period and subject; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of (-2, 2). A prespecified equivalence margin of (-2,2) was used for equivalence analysis; Mean Difference (Final Values) = 0.1, 95% CI [-0.09 to 0.28], Standard Error of Mean 0.09

2. Secondary Outcome: The Number of Patients Requiring Rescue Medication During the DB Tapentadol IR Treatment
Time Frame: 14 days for each cross-over period
Population: DB safety set defined as randomized subjects who took at least one dose of study drug during the DB treatment period.
Measure: Number; unit: participants
Arm/Group | Tapentadol
Number analyzed (Participants) | 81
participants | 24

3. Secondary Outcome: The Number of Patients Requiring Rescue Medication During the DB Tapentadol ER Treatment
Time Frame: 14 days for each cross-over period
Population: DB safety set defined as randomized subjects who took at least one dose of study drug during the DB treatment period.
Measure: Number; unit: participants
Arm/Group | Tapentadol
Number analyzed (Participants) | 84
participants | 29

4. Secondary Outcome: Total Daily Dose (TDD) of Tapentadol IR During the Double-blind Treatment Period
Description: Average total daily dose (TDD) of tapentadol IR during the double blind treatment period
Time Frame: 14-day for each DB treatment period
Population: DB safety set defined as randomized subjects who took at least one dose of study drug during the DB treatment period.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Tapentadol
Number analyzed (Participants) | 81
mg | 331.0 (116.17)

5. Secondary Outcome: Total Daily Dose (TDD) of Tapentadol ER During the DB Treatment Period.
Description: Average total daily dose (TDD) of tapentadol ER during the double-blind treatment period.
Time Frame: 14 days for each treatment period
Population: DB safety set defined as randomized subjects who took at least one dose of study drug during the DB treatment period.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Tapentadol
Number analyzed (Participants) | 84
mg | 330.4 (123.73)

ADVERSE EVENTS:
Time Frame: All adverse events were reported from the time a signed and dated informed consent was obtained throughout the follow-up phase of the study (up to 63 days post dose). Serious adverse events were collected for 30 days after the last dose of study drug.
Groups:
- Tapentadol: Subjects treated in the Tapentadol Immediate Release (IR) open-label and the double-blind crossover period.
Arm/Group | Tapentadol
Serious Adverse Events (participants affected / at risk) | 2/116
Other Adverse Events (participants affected / at risk) | 98/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tapentadol (N=116)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol (N=116)
Dizziness (Nervous system disorders) | 28
Headache (Nervous system disorders) | 19
Somnolence (Nervous system disorders) | 19
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 8
Dry Mouth (Gastrointestinal disorders) | 6
Upper Respiratory Tract Infection (Infections and infestations) | 9
Fatigue (General disorders) | 10
Pyrexia (General disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 9
Anxiety (Psychiatric disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days